CLINICAL TRIAL: NCT03441256
Title: Motor, Sensory, and Autonomic Function After Laparoscopic Implantation of Neuroprosthesis - a Randomized Controlled Trial of the LION Procedure in Traumatic Spinal Cord Injury
Brief Title: Motor, Sensory, and Autonomic Function in Traumatic Spinal Cord Injury After the LION Procedure.
Acronym: SCI-LION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spinal Cord Injury Centre of Western Denmark (Other)
Collaborators: Aarhus University Hospital (Other); Regionshospitalet Viborg, Skive (Other); University of Southern Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VCR-SBE-01
Record Dates: First submitted 2018-01-24; First posted 2018-02-22 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-03

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): All participant in the intervention group will undergo the LION procedure and subsequent neurostimulation.
  Interventions: Device: LION procedure
- Control (Active Comparator): All participants in the control group will be issued with a device for neuromuscular electrical stimulation.
  Interventions: Device: NMES

INTERVENTIONS:
Device: LION procedure — Laparoscopic implantation of an impulse generator and four leads for electrical stimulation of femoral and sciatic nerves.
  Other Names: Neurostimulation
  Arms: Intervention
Device: NMES — Conventional neuromuscular electrical stimulation via surface electrodes.
  Other Names: Neuromuscular electrical stimulation
  Arms: Control

SUMMARY:
Possover pioneered a minimally invasive and fully reversible laparoscopic technique, laparoscopic implantation of neuroprosthesis (LION), for precise placement of an implantable pulse generator and one to four leads for stimulating nerves of the lumbosacral plexus.

Unexpectedly, Possover in 2014 made the clinical observation that four patients with complete and incomplete chronic traumatic spinal cord injury regained significant motor and sensory function following the LION procedure for bladder and bowel dysfunction.

The primary objective of this randomized clinical trial is to investigate whether the LION procedure and the subsequent neurostimulation in individuals with chronic traumatic thoracolumbar spinal cord injury with spastic paraplegia is associated with increased walking capacity.

DETAILED DESCRIPTION:
Sustaining a spinal cord injury impacts the mental and physical wellbeing of the injured individuals profoundly; quality of life suffers and subsequently the risk of suicide is greatly increased as compared to the general population. While spinal cord injury compromises an individual's mobility, dependency does not necessarily ensue; most individuals will require a wheelchair, braces or other assistive devices for maintaining activities of daily living and participating in society i.e. work, sport etc.

Furthermore, individuals with spinal cord injury face numerous medical complications and reduced life expectancy as a direct result of their disability.Detrusor over-activity and sphincter dyssynergia are seen in up to 85% of cases and improved control of micturition and defaecation closely follows restoration of ambulation as primary rehabilitation goals of patients with spinal cord injury.

Recovery after initial inpatient rehabilitation is at best modest and conversion rate of the American Spinal Injury Association Impairment Scale grade remain poor for grades A and B. Likewise, the rate of motor improvement stagnates over time leaving many patients with permanent motor, sensory and autonomic deficits. 9-12 months after their initial injury, most patients have essentially exhausted their possibility of further restorative treatments.

Possover pioneered a minimally invasive and fully reversible laparoscopic technique, laparoscopic implantation of neuroprosthesis (LION), for precise placement of an implantable pulse generator and one to four leads for stimulating nerves of the lumbosacral plexus; a significant number cases suggest this technique is safe and efficacious in treating overactive and atonic bladder disturbances, neurogenic bowel dysfunction, and abdominopelvic neuropathic pain.

Unexpectedly, Possover in 2014 made the clinical observation that four patients with complete and incomplete chronic traumatic spinal cord injury regained significant motor and sensory function following the LION procedure for bladder and bowel dysfunction. Expanding further on the topic, Possover have recently published an updated case series of 18 patients om whom 16 are now capable of weight bearing standing and 12 are furthermore capable of voluntary stepping.

The primary objective of this randomized clinical trial is therefore to investigate whether the LION procedure and the subsequent neurostimulation in individuals with chronic traumatic thoracolumbar spinal cord injury with spastic paraplegia is associated with increased walking capacity.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to give informed consent for participation in the clinical investigation, and to comply with all requirements of the clinical investigation
2. Traumatic SCI with:

   * neurological level below T5 and above L2
   * American Spinal Injury Association Impairment Grade A or B
   * spasticity in one or both lower extremities
   * Injury prior at least 12 months prior to enrollment

Exclusion Criteria:

1. Female subject who is pregnant/planning pregnancy during the clinical investigation.
2. Previous surgery/procedures interfering with the LION procedure incl. the presence of other implanted medical devices.
3. Any other significant disease or disorder which, in the opinion of the Investigator, may either put the subject at risk because of participation in the clinical investigation, or may influence the result of the clinical investigation, or the subject's ability to participate in the clinical investigation

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Improvement/change in walking capacity | Baseline, 3 mo., 6 mo., 9 mo., 12 mo.
  Walking index for spinal cord injury, second revision (WISCI II)

SECONDARY OUTCOMES:
Change in lean body mass | Baseline, 12 mo.
  Changes in lean body mass on dual-energy x-ray absorptiometry
Change in distal motor latency of motor nerve conduction studies | Baseline, 12 mo.
  Preoperative to postoperative change in distal motor latency of the compound muscle action potential.
Change in peak-peak amplitude of motor nerve conduction studies | Baseline, 12 mo.
  Preoperative to postoperative change in change in peak to peak amplitude of the compound muscle action potential.
Change in muscle microarchitecture | Baseline, 12 mo.
  Preoperative to postoperative changes in fiber-type composition on histochemical analysis of soles muscle biopsies.
Change in muscle motor unit number | Baseline, 12 mo.
  Preoperative to postoperative changes in motor unit number estimation.
Change in compound muscle action potential scans. | Baseline, 12 mo.
  Preoperative to postoperative changes in compound muscle action potential scan slope.
Change in sensory nerve action potential latency of sensory nerve conduction studies | Baseline, 12 mo.
  Preoperative to postoperative change in sensory nerve action potential latency.
Change in peak-peak amplitude of the sensory nerve action potential of sensory nerve conduction studies | Baseline, 12 mo.
  Preoperative to postoperative change in peak-peak amplitude of the sensory nerve action potential.
Change in sensory discrimination | Baseline, 12 mo.
  Change in parameters of quantitative sensory testing applying method of limits.
Change in bowel function | Baseline, 12 mo.
  Changes in scores on the international spinal cord injury data set - bowel function
Change in bladder function | Baseline, 12 mo.
  Changes in scores on the international spinal cord injury data set - lower urinary tract function
Change in health-related quality of life | Baseline, 12 mo.
  Changes in scores of the international spinal cord injury data set - quality of life
Change in quality of life | Baseline, 12 mo.
  Changes in the scores of the Short Form 36 questionnaire; the questionnaire has eight subscales (vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, and mental health). Each sub scale scores 0-100, 0 indicating maximal disability.
Change in pain | Baseline, 3 mo., 6 mo., 9 mo., 12 mo.
  Changes in the brief pain inventory questionnaire; questionnaire consists of 17-items addressing pain severity, pain location, pain chronicity, and amount of pain relief. Each item scores are 0-10, 10 indicating either maximum pain severity, maximum interference or maximum relief, respectively.
Change in spasticity | Baseline, 12 mo.
  Changes in scores of the modified Tardieu Scale for spasticity; scores 0-4, 4 being maximum level of spasticity.

CONTACTS AND LOCATIONS:
Overall Officials: Helge Kasch, MD, Study Director — Spinal Cord Injury Centre of Western Denmark
Locations (1):
- Helge Kasch, Viborg, Central Jutland, Denmark

IPD SHARING:
Plan to Share IPD: No
Individual participant data may be requested by other researchers. Approvals from the Danish Data Protection Agency and individual participants will be required before data may be shared.

REFERENCES:
- [Derived] Possover M, Abrao HM. Low-frequency antidromic pelvic neuromodulation as a potential enhancer of recovery after spinal cord injury: hypothetical promotion of spinal Renshaw cells and corticovagal plasticity. J Spinal Cord Med. 2025 Sep 15:1-7. doi: 10.1080/10790268.2024.2414146. Online ahead of print. PMID 40952735
- See also: Effect of pelvic laparoscopic implantation of neuroprosthesis in spinal cord injured subjects: a 1-year prospective randomized controlled study — http://www.nature.com/articles/s41393-021-00693-7
- See also: Surgical Aspects of the Possover LION Procedure: An Emerging Procedure for Recovery of Visceral Functions and Locomotion in Paraplegics — http://doi.org/10.5005/jp-journals-10033-1450